CLINICAL TRIAL: NCT01321398
Title: Transpulmonary Pressure Gradients in High Frequency Oscillation Study
Brief Title: Transpulmonary Pressure Gradients in High Frequency Oscillation
Acronym: TPG in HFO
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H10-02087
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Acute Lung Injury
Keywords: High Frequency Oscillation; Oscillation; HFO; Transpulmonary pressure
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Critically Ill patients receiving HFO
  Interventions: Other: Esophageal Pressure Monitoring

INTERVENTIONS:
Other: Esophageal Pressure Monitoring — An esophageal pressure monitor will be placed through the mouth into the esophagus by a study physician. Placement will be confirmed by a bedside chest X-ray. Once placement has been confirmed all air will be evacuated from the balloon by syringe. One ml of air will then be injected to partially inflate the esophageal balloon. Pleural pressure measurements will be recorded after 1 minute without spontaneous breathing or patient care related movement. This measurement will be repeated at 30 minutes and at 60 minutes after the first measurement. Trans-pulmonary pressure is calculated as the difference between esophageal pressure and mouth pressure. Once the measurements have been recorded, the catheter will be removed.

SUMMARY:
Patients with severe lung conditions occasionally require support with a special ventilator (breathing machine) called the High Frequency Oscillator (HFO). Effective ventilation requires that the pressure generated by the ventilator be as high as possible but not too high as this can damage the lungs. In patients on HFO, there is not a well defined way to measure this pressure. We will insert a small probe into the esophagus of patients on HFO to see if this is an accurate way to measure lung pressures for these patients. A better understanding of these pressures could lead to improved patient care.

DETAILED DESCRIPTION:
Trials have found that the use of lower tidal volumes (6 ml/kg) during conventional mechanical ventilation decreases morbidity and mortality. Compared to conventional ventilation, high frequency oscillation (HFO) is able to provide much smaller tidal volumes (1.1 - 2.5 ml/kg) and thus theoretically may provide additional lung protection. At this time, while trials of HFO in adults have been inconclusive, the use of HFO for the management of ALI/ARDS has become widespread

Patients with acute lung injury (ALI) or acute respiratory distress syndrome (ARDS) are critically ill and have a high mortality associated with their illness (approximately 50%). Currently, esophageal pressure monitors are used to optimize inflation pressures and improve oxygenation in conventional mechanical ventilation in patients with ALI/ARDS. With this in mind, the purpose of this study is twofold: (1) demonstrate that esophageal pressure monitors can easily be inserted in patients undergoing HFO and (2) report the transpulmonary pressures in these patients.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* Receiving HFO
* Informed Consent Obtained

Exclusion Criteria:

* Esophageal lesions or esophageal surgery within the last 6 months
* Morbid obesity - defined as a Body Mass Index (BMI) > 40
* Unstable cervical spine injury or cervical spinal cord injury

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically Ill
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To demonstrate the proof of concept that esophageal pressures can easily be obtained in patients undergoing HFO. | 60 minutes

SECONDARY OUTCOMES:
To determine the transpulmonary pressure gradient in critically ill patients receiving HFO | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: William R Henderson, FRCPC, Principal Investigator — Universtiy of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada